CLINICAL TRIAL: NCT00697008
Title: Symptomatic Assessment and Therapeutic Outcomes in Typical GERD Patients Following a New CP Guideline in the Clinical Practice
Brief Title: Asociación Española de Gastroenterologia (Spanish Gastroenterology Association) Gastroesophageal Reflux Disease Guideline - Prospective Study
Acronym: Prospect
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Mercedes Muñoz, PhD, Local MC GI Therapeutic Area Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GES-DUM-2007/3
Record Dates: First submitted 2008-06-04; First posted 2008-06-13 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: GERD
Keywords: GERD; CLINICAL GUIDELINE; Symptoms; clinical outcome
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GERD patients: Patients with typical GERD symptoms

SUMMARY:
To evaluate symptomatic outcome and HRQoL in GERD patients treated following a new CP Guideline.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age above 18
* Subjects with typical GERD symptoms: predominant heartburn/regurgitation
* Naive patients or off PPI treatment in the last 2 months

Exclusion Criteria:

* Inability to read and understand PRO instructions
* Patient not suitable to be treated following the AEG guidelines
* Concomitant treatment with NSAID, antiplatelet drugs
* Previous PPI failure

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with typical GERD symptoms consulting in specialized care setting and are managed following the new local GERD guidelines
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Symptomatic outcome of GERD management following new guideline | End of study visit 4-8w

SECONDARY OUTCOMES:
To evaluate the frequency and type of extraesophageal and dyspeptic symptoms and their impact on the clinical outcome | End of study 4-8w
To evaluate the impact of GERD symptoms in HRQoL | End of study 4-8w

CONTACTS AND LOCATIONS:
Overall Officials: Javier Zapardiel, MD, Study Chair — AZ SPAIN
Locations (29):
- Spain (29):
  - Research Site, Badajoz, Badajoz
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Barcelona, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Viladecans, Barcelona
  - Research Site, Cadiz, Cadiz
  - Research Site, Jerez de la Frontera, Cadiz
  - Research Site, Cabra, Cordoba
  - Research Site, Córdoba, Cordoba
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Huelva, Huelva
  - Research Site, Huesca, Huesca
  - Research Site, A Coruña, La Coruna
  - Research Site, Santiago de Compostela, La Coru�a
  - Research Site, Madrid, Madrid
  - Research Site, Marbella, Malaga
  - Research Site, Málaga, Malaga
  - Research Site, Murcia, Murcia
  - Research Site, Verín, Orense
  - Research Site, Vigo, Pontevedra
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Seville, Sevilla
  - Research Site, Tarragona, Tarragona
  - Research Site, LA Cuesta de Arguijon, Tenerife
  - Research Site, Alzira, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Barakaldo, Vizcaya
  - Research Site, Bilbao, Vizcaya
  - Research Site, Zaragoza, Zaragoza